CLINICAL TRIAL: NCT01634412
Title: A Single-Dose, Open-Label, Randomized Study of the Comparative Pharmacokinetics of Sublingual TNX-102 2.4 mg at pH 3.5 and 7.1, Oral Cyclobenzaprine 5 mg Tablets, and Intravenous Cyclobenzaprine 2.4 mg in Healthy Adults
Brief Title: Comparative Bioavailability of Sublingual TNX-102, Oral and Intravenous Cyclobenzaprine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tonix Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TNX-CY-F102
Record Dates: First submitted 2012-06-25; First posted 2012-07-06 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Healthy Adults
MeSH Terms: interventions — cyclobenzaprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- SL TNX-102 at pH 3.5 (Experimental): 2.4 mg TNX-102 sublingual solution (2.4 mg/mL) in PBS at pH 3.5
  Interventions: Drug: SL TNX-102 2.4 mg at pH 3.5
- SL TNX-102 at pH 7.1 (Experimental): 2.4 mg TNX-102 sublingual solution (2.4 mg/mL) in PBS at pH 7.1
  Interventions: Drug: SL TNX-102 2.4 mg at pH 7.1
- Cyclobenzaprine tablets (Active Comparator): 5 mg cyclobenzaprine tablet once
  Interventions: Drug: Cyclobenzaprine Tablet
- Cyclobenzaprine IV (Active Comparator): 2.4 mg cyclobenzaprine USP in PBS (0.6 mg/mL) at pH 7.4
  Interventions: Drug: Cyclobenzaprine IV

INTERVENTIONS:
Drug: SL TNX-102 2.4 mg at pH 3.5 — 1 dose of 2.4 mg TNX-102 sublingual solution (2.4 mg/mL) in PBS at pH 3.5, administered as 1 mL held under the tongue for 90 seconds without swallowing
  Arms: SL TNX-102 at pH 3.5
Drug: SL TNX-102 2.4 mg at pH 7.1 — 1 dose of 2.4 mg TNX-102 sublingual solution (2.4 mg/mL) in PBS at pH 7.1, administered as 1 mL held under the tongue for 90 seconds without swallowing
  Arms: SL TNX-102 at pH 7.1
Drug: Cyclobenzaprine Tablet — 1 x 5 mg cyclobenzaprine tablet, swallowed with 240 mL of room-temperature water
  Arms: Cyclobenzaprine tablets
Drug: Cyclobenzaprine IV — 1 dose of 2.4 mg cyclobenzaprine USP in PBS (0.6 mg/mL) at pH 7.4, administered intravenously as a 4 mL bolus injection over 30 seconds
  Arms: Cyclobenzaprine IV

SUMMARY:
Very low dose (VLD) cyclobenzaprine at bedtime has shown promise as a treatment for fibromyalgia, but the chemistry of cyclobenzaprine requires new formulation technology for bedtime use. The present trial is designed to assess the safety and tolerability of sublingual TNX-102 2.4 mg (a new formulation of cyclobenzaprine designed to result in increased dosage precision and decreased potential for morning grogginess) at pH 3.5 and 7.1 and to compare the bio-availability of sublingual TNX-102 2.4 mg at pH 3.5 and 7.1 and cyclobenzaprine (5 mg tablets, or 2.4 mg iv).

ELIGIBILITY:
Inclusion Criteria: Healthy adults

* Male or female
* Non-smoker
* 18-65 years old
* BMI > 18.5 and < 30.0
* With medically acceptable form of contraception (female only)
* With signed informed consent

Exclusion Criteria:

* Any clinically significant abnormality including ECG abnormalities or vital sign abnormalities (systolic blood pressure < 90 or > 140 mmHg, diastolic blood pressure lower < 50 or > 90 mmHg, or heart rate < 50 or > 100 BPM)
* Any abnormal laboratory test (including positivity for Hep B, Hep C, HIV, and Hemoglobin < 128 g/L (males) or < 115 g/L (females) and hematocrit < 0.37 L/L (males) or < 0.32 L/L (females))
* History of alcohol or drug abuse or dependence within 1 year and/or positive drug, cotinine, or alcohol tests
* Use of any drug (within 30 days), supplement, or food (within 14 days) known to induce or inhibit hepatic drug metabolism prior to study medication
* Positive pregnancy test, breastfeeding or lactating
* Use of medication other than hormonal contraceptives or topical products, including OTC, natural health products, MAO inhibitors
* Participation in an investigational study within 30 days prior to dosing
* Donation of plasma (within 7 days), or donation or loss of blood of 50-499 mL (within30 days), or of > 499 mL (within 56 days) prior to dosing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-06; Primary Completion 2013-09 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
• Measured levels of cyclobenzaprine and norcyclobenzaprine in plasma and urine | 27 time points per period for blood assessment ; 3 pooled analyses in urine.
  Blood samples will be taken per period: within 30 minutes pre-dose and 2, 3.5, 5, 10, 20, 30, and 45 minutes and 1, 2, 2.5, 3, 3.33, 3.67, 4, 4.33, 4.67, 5, 5.5, 6, 8, 12, 16, 24, 36, 48, and 72 hours post-dose. A single urine sample will be collected within 30 minutes pre-dose (one sample), and urine will be pooled from 0-24, 24-48 and 48-72 hours post-dose.
Safety and tolerability of sublingual TNX-102 2.4 mg at pH 3.5 and pH 7.1. | Continuously until the end (day 4) of the study period + Telephone follow-up 7-13 days after dosing (total duration: about 1 month)
  Every adverse events occurring during the study period will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Seth M. Lederman, MD, Study Chair — Tonix Pharmaceuticals, Inc.; Jeffrey P. Kitrelle, MD, Study Director — Tonix Pharmaceuticals, Inc.; Denis Audet, MD, Principal Investigator — PharmaNet
Locations (1):
- PharmaNet, Inc., Québec, Quebec, Canada